CLINICAL TRIAL: NCT01241435
Title: The Effect of Impaired Hepatic Function on the Pharmacokinetics of LY2216684
Brief Title: A Study of LY2216684 in Participants With Impaired Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12602; H9P-EW-LNCM (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-11-12; First posted 2010-11-16 (Estimated); Results first posted 2018-10-22 (Actual); Last update posted 2018-10-22 (Actual); Status verified 2018-03

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — alpha-((5-fluoro-2-methoxyphenyl)methyl)-alpha-(tetrahydro-2H-pyran-4-yl)-2-morpholinemethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LY2216684 (Experimental): LY2216684: A single dose of 18 milligrams (mg) administered orally in participants with normal hepatic function, mild hepatic impairment (Child-Pugh A), moderate hepatic impairment (Child-Pugh B), or severe hepatic impairment (Child-Pugh C)
  Interventions: Drug: LY2216684

INTERVENTIONS:
Drug: LY2216684 — Administered orally
  Other Names: Edivoxetine

SUMMARY:
The purpose of this study is to evaluate the effect of liver function on how much of the study drug (LY2216684) gets into the blood stream and how long it takes the body to get rid of it. Information about any side effects that may occur will also be collected.

The duration of participation in this study is approximately 12 days, not including the screening visit. This study requires 1 clinic confinement of 5 days/4 nights followed by 1 out-patient follow-up visit. A screening visit is required within 30 days prior to the start of the study. This research study will be an open-label study.

The study involves a single oral dose of 18 milligrams (mg) LY2216684 given as 2 tablets.

ELIGIBILITY:
Inclusion Criteria:

* Male participants: Agree to use a reliable method of birth control during the study and for 3 months following the last dose of study drug.
* Female participants: Are women of child-bearing potential who test negative for pregnancy at the time of enrollment, who have used a reliable method of birth control for 6 weeks prior to administration of study drug, and who agree to use a reliable method of birth control during the study and for 1 month following the last dose of study drug or are women not of child-bearing potential due to surgical sterilization (hysterectomy, bilateral oophorectomy, or tubal ligation) or menopause (at least 1 year without menses or 6 months without menses and follicle stimulating hormone [FSH] levels greater than or equal to 40 milli-internation units per milliliter [mIU/mL]).
* Have a body mass index (BMI) of 17.0 to 35.0 kilograms per meters squared (kg/m^2), inclusive, at screening.
* Have acceptable blood pressure and pulse rate (sitting) as determined by the investigator.
* Have venous access sufficient to allow blood sampling as per the protocol.
* Are reliable and willing to make themselves available for the duration of the study and to follow study procedures.
* Have given written informed consent approved by Lilly and the institutional review board (IRB) governing the site.

Control Participants (Participants with Normal Hepatic Function):

* Are overtly healthy, as determined by medical history and physical examination.
* Have clinical laboratory test results within normal reference ranges for the investigative site or results with acceptable deviations, which are judged to be not clinically significant by the investigator, at the time of screening.

Participants with Mild, Moderate, or Severe Hepatic Impairment:

* Participants with stable liver disease (alcoholic liver disease, post-hepatitis, biliary cirrhosis, cryptogenic) classified as Child-Pugh score A, B, or C (Pugh et al. 1973).
* Clinical laboratory test results with deviations that are judged by the investigator to be compatible with the hepatic impairment of the participant or of no additional clinical significance for this study.

Exclusion Criteria:

All Participants:

* Are currently enrolled in, or discontinued within the last 30 days from a clinical trial involving an investigational drug or device or off-label use of a drug or device other than the study drug used in this study or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
* Have known allergies to LY2216684 or related compounds.
* Are persons who have previously completed or withdrawn from this study or any other study investigating LY2216684 in the past 6 months from screening.
* Have an electrocardiogram (ECG) reading considered clinically significant by the investigator or a history of significant cardiac dysrhythmia or conduction defect that, in the opinion of the investigator, increases the risks associated with participating in the study.
* Show evidence of human immunodeficiency virus (HIV) and/or positive human HIV antibodies.
* There is evidence or history of neurological disease such as transient ischemic attack, stroke, syncope episodes, encephalitis, or meningitis, except participants with liver disease-related encephalopathy may be allowed.
* Presence of acute infection with fever.
* Are women with a positive pregnancy test or women who are lactating.
* Have lost 500 milliliters (mL) or more of blood in the 3 months prior to study entry.
* Are participants who have an average weekly alcohol intake that exceeds 21 units per week, or are unwilling to adhere to restrictions during the study (1 unit = 12 ounces [oz] or 360 mL of beer, 5 oz or 150 mL of wine, or 1.5 oz or 45 mL of distilled spirits).
* Are participants who are unwilling to adhere to study caffeine restrictions.
* Are participants who are unwilling to abide by smoking restrictions while resident in the clinical research unit (CRU).
* Have a documented or suspected history of glaucoma.

Control Participants (Participants with Normal Hepatic Function):

* Have significant active hematological disease, history of significant active bleeding, or coagulation disorder.
* Use or intend to use over-the-counter (including vitamins/mineral supplements, herbal medicine) or prescription medications 14 days, prior to enrollment and during the study.
* Have history or presence of cardiovascular, respiratory, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data.
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening.
* Evidence of hepatitis C and/or positive hepatitis C antibody.
* Evidence of hepatitis B and/or positive hepatitis B surface antigen.
* Show evidence of significant active neuropsychiatric disease.

Participants with Mild, Moderate, or Severe Hepatic Impairment:

* Evidence of any significant active disease other than that responsible for or associated with liver impairment.
* Have history or presence of cardiovascular, respiratory, renal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs or of constituting a risk when taking the study medication or interfering with the interpretation of data.
* Evidence of hepatorenal syndrome.
* Spontaneous bacterial peritonitis within 6 months of study entry.
* Variceal bleeding within 3 months of study entry.
* Severe hyponatremia (sodium [Na] <120 millimole per liter [mmol/L]).
* Presence of hepatocellular carcinoma.
* Severe encephalopathy.
* Hemoglobin <9.0 grams per deciliter (g/dL).
* Platelet count <50 x 10^9 cells per liter (cells/L), values <50 x 10^9 cells/L may be permitted at the discretion of the investigator in consultation with the sponsor.
* Concomitant use of any drug except those indicated for the treatment of liver disease or related complications.
* Concomitant use of anticoagulants including warfarin.
* Regular use of drugs of abuse and/or positive findings on urinary drug screening except those prescribed for related complications (such as, pain, insomnia, or anxiety) of liver disease.
* The use of medication known to interfere with hepatic metabolism (such as, barbiturates or phenothiazines) or known to alter other major organs or systems within 30 days prior to study entry.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-10; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Normal Hepatic Function: LY2216684: A single dose of 18 milligrams (mg) administered orally in participants with normal hepatic function
- Mild Hepatic Impairment: LY2216684: A single dose of 18 milligrams (mg) administered orally in participants with mild hepatic impairment (Child-Pugh A)
- Moderate Hepatic Impairment: LY2216684: A single dose of 18 milligrams (mg) administered orally in participants with moderate hepatic impairment (Child-Pugh B)
- Severe Hepatic Impairment: LY2216684: A single dose of 18 milligrams (mg) administered orally in participants with severe hepatic impairment (Child-Pugh C)
Period: Overall Study
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Started | 12 | 8 | 8 | 8
Received at Least 1 Dose of Study Drug | 12 | 8 | 8 | 8
Completed | 12 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment | Total
Number analyzed (Participants) | 12 | 8 | 8 | 8 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (6.3) | 55.0 (4.9) | 54.5 (5.6) | 51.4 (6.9) | 52.3 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 2 | 1 | 10
  Male | 8 | 5 | 6 | 7 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 10 | 8 | 8 | 8 | 34
  Black/African American | 1 | 0 | 0 | 0 | 1
  Multiple | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 8 | 8 | 8 | 36

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Area Under the Concentration Curve (AUC)
Description: The area under the plasma concentration versus time curve from 0 hours to infinity (AUC [0-∞]) for LY2216684 is presented.
Time Frame: Up to 72 hours after administration of study drug
Population: Participants who received at least one dose of study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours times nanograms/milliliter
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 12 | 8 | 8 | 8
hours times nanograms/milliliter | 601 (32) [503 to 717] | 742 (52) [598 to 922] | 961 (45) [774 to 1194] | 1020 (16) [820 to 1265]

2. Primary Outcome: Pharmacokinetics: Maximum Concentration (Cmax)
Time Frame: Up to 72 hours after administration of study drug
Population: Participants who received at least one dose of study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 12 | 8 | 8 | 8
nanograms/milliliter | 46.8 (27) | 39.6 (28) | 41.9 (33) | 34.7 (15)

3. Primary Outcome: Pharmacokinetics: Time to Maximum Concentration (Tmax)
Time Frame: Up to 72 hours after administration of study drug
Population: Participants who received at least one dose of study drug.
Measure: Median (Full Range); unit: hours
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Number analyzed (Participants) | 12 | 8 | 8 | 8
hours | 3.00 [1.00 to 5.00] | 3.50 [2.00 to 6.00] | 3.50 [1.00 to 5.00] | 3.50 [2.00 to 5.00]

ADVERSE EVENTS:
Arm/Group | Normal Hepatic Function | Mild Hepatic Impairment | Moderate Hepatic Impairment | Severe Hepatic Impairment
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 6/12 | 3/8 | 6/8 | 5/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Normal Hepatic Function (N=12) | Mild Hepatic Impairment (N=8) | Moderate Hepatic Impairment (N=8) | Severe Hepatic Impairment (N=8)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1) | 2 (2)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary hesitation (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days